CLINICAL TRIAL: NCT01063829
Title: A Randomized, Double-blind, Placebo Controlled Trial to Evaluate the Safety, Tolerability and Antiviral Activity of 12 Weeks' Treatment With a New Antiviral HCMV Drug
Brief Title: Safety and Efficacy Study of a New Antiviral Drug to Prevent Cytomegalovirus Reactivation in Bone Marrow Transplanted Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AiCuris Anti-infective Cures AG (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AIC246-01-II-02
Record Dates: First submitted 2010-02-04; First posted 2010-02-05 (Estimated); Results first posted 2018-02-13 (Actual); Last update posted 2018-02-13 (Actual); Status verified 2010-12

CONDITIONS: HCMV Reactivation or HCMV End-Organ Disease
Keywords: HCMV
MeSH Terms: interventions — letermovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Dose regimen 1 (Experimental): 60 mg AIC246, one tablet per day
  Interventions: Drug: 60 mg AIC246
- Dose regimen 2 (Experimental): 120 mg AIC246, one tablet per day
  Interventions: Drug: 120 mg AIC246
- Dose regimen 3 (Experimental): 240 mg AIC246, one tablet per day
  Interventions: Drug: 240 mg AIC246
- Placebo (Other): Placebo arm
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: 60 mg AIC246 — Oral administration
  Arms: Dose regimen 1
Drug: 120 mg AIC246 — Oral administration
  Arms: Dose regimen 2
Drug: 240 mg AIC246 — Oral administration
  Arms: Dose regimen 3
Other: Placebo — Oral administration
  Arms: Placebo

SUMMARY:
The aim of the study is to find out whether AIC246 is safe and efficacious in lowering the chances of the cytomegalovirus becoming active again and causing illness after an HBPC transplant (allogeneic stem cell transplant).

ELIGIBILITY:
Inclusion Criteria:

* Seropositive for HCMV IgG antibodies before transplantation
* First allogeneic Human blood precursor cell (HBPC) transplantation performed for 1 of the following diagnoses: leukaemia, lymphoma, Hodgkin's lymphoma, non-Hodgkin's lymphoma, multiple myeloma, myelodysplastic and myeloproliferative disorder
* Evidence of post transplantation engraftment
* Able to swallow tablets.

Exclusion Criteria:

* Previous anti-HCMV therapy after this allogeneic HBPC transplantation
* Mismatched or cord blood transplant recipients
* Current or history of end-organ HCMV disease
* Graft versus host disease (GVHD)
* Impaired liver function
* Reduced renal function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2010-03; Primary Completion 2011-10 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (24):
- United States (14):
  - UCLA Medical Center, Los Angeles, California
  - Stanford University Hospital, Stanford, California
  - Denver St. Lukes Presbyterian, Denver, Colorado
  - University of Florida, Gainesville, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - Loyola University Chicago, Maywood, Illinois
  - Indiana BMT, Beech Grove, Indiana
  - University Of Iowa, Iowa City, Iowa
  - Dana Farber Cancer Institute,, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Jeanes Hospital of TUHS, Philadelphia, Pennsylvania
  - UPMC Cancer Center, Pittsburgh, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
- Germany (10):
  - Universitaetsklinikum Dresden, Dresden
  - Universitaetsklinikum Erlangen-PS, Erlangen
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
  - Universitaeetsklinikum Heidelberg, ,, Heidelberg
  - Universitaetsklinikum Mainz, Mainz
  - Universitaetsklinikum Muenster, Münster
  - Klinikum Nuernberg Nord, Nuremberg
  - Robert-Bosch-Krankenhaus, Stuttgart
  - Universitaetsklinikum Wuerzburg, Würzburg

REFERENCES:
- [Derived] Chemaly RF, Ullmann AJ, Stoelben S, Richard MP, Bornhauser M, Groth C, Einsele H, Silverman M, Mullane KM, Brown J, Nowak H, Kolling K, Stobernack HP, Lischka P, Zimmermann H, Rubsamen-Schaeff H, Champlin RE, Ehninger G; AIC246 Study Team. Letermovir for cytomegalovirus prophylaxis in hematopoietic-cell transplantation. N Engl J Med. 2014 May 8;370(19):1781-9. doi: 10.1056/NEJMoa1309533. PMID 24806159

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 133 patients were randomized to the trial; 2 randomized patients did not receive the assigned study drug ( 1 Patient died and 1 Patient had CMV reactivation before intended administartion of first dose)
Groups:
- AIC246 (60 mg); AIC246 (120 mg); AIC246 (240 mg): AIC246: Oral Administration
Period: Overall Study
Arm/Group | AIC246 (60 mg) | AIC246 (120 mg) | AIC246 (240 mg) | Placebo
Started | 33 | 31 | 34 | 33
Completed | 17 (Non-completers considered as failure; FAS) | 21 (Non-completers considered as failure; FAS) | 24 (Non-completers considered as failure; FAS) | 12 (Non-completers considered as failure; FAS)
Not Completed | 16 | 10 | 10 | 21

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AIC246 (60 mg) | AIC246 (120 mg) | AIC246 (240 mg) | Placebo | Total
Number analyzed (Participants) | 33 | 31 | 34 | 33 | 131
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.5 (13.03) | 51.6 (12.79) | 50.7 (11.78) | 51.8 (13.41) | 51.1 (12.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 9 | 12 | 14 | 54
  Male | 14 | 22 | 22 | 19 | 77
Region of Enrollment [Number; unit: participants]
  United States | 18 | 19 | 17 | 15 | 69
  Germany | 15 | 12 | 17 | 18 | 62

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With "HCMV Prophylaxis Failure"
Time Frame: 84 days
Measure: Count of Participants; unit: Participants
Arm/Group | AIC246 (60 mg) | AIC246 (120 mg) | AIC246 (240 mg) | Placebo
Number analyzed (Participants) | 33 | 31 | 34 | 33
Participants | 16 | 10 | 10 | 21
Statistical Analysis 1: Comparison: AIC246 (240 mg) vs Placebo; Test type: Superiority or Other; p = 0.007, Fisher Exact
Statistical Analysis 2: Comparison: AIC246 (120 mg) vs Placebo; Test type: Superiority or Other; p = 0.014, Fisher Exact
Statistical Analysis 3: Comparison: AIC246 (60 mg) vs Placebo; Test type: Superiority or Other; p = 0.321, Fisher Exact

2. Primary Outcome: Time to Onset of "HCMV Prophylaxis Failure"
Time Frame: 84 days
Measure: Number; unit: days
Arm/Group | AIC246 (60 mg) | AIC246 (120 mg) | AIC246 (240 mg) | Placebo
Number analyzed (Participants) | 33 | 31 | 34 | 33
days | 7 | 6 | 2 | 12
Statistical Analysis 1: Comparison: AIC246 (240 mg) vs Placebo; Test type: Superiority or Other; p = 0.002, Log Rank
Statistical Analysis 2: Comparison: AIC246 (120 mg) vs Placebo; Test type: Superiority or Other; p = 0.126, Log Rank
Statistical Analysis 3: Comparison: AIC246 (60 mg) vs Placebo; Test type: Superiority or Other; p = 0.148, Log Rank

3. Secondary Outcome: Number of Patients With Systemic Detectable HCMV Replication.
Time Frame: 84 days
Measure: Count of Participants; unit: Participants
Arm/Group | AIC246 (60 mg) | AIC246 (120 mg) | AIC246 (240 mg) | Placebo
Number analyzed (Participants) | 33 | 31 | 34 | 33
Participants | 7 | 5 | 2 | 12
Statistical Analysis 1: Comparison: AIC246 (240 mg) vs Placebo; Test type: Superiority or Other; p = 0.007, Fisher Exact
Statistical Analysis 2: Comparison: AIC246 (120 mg) vs Placebo; Test type: Superiority or Other; p = 0.014, Fisher Exact
Statistical Analysis 3: Comparison: AIC246 (60 mg) vs Placebo; Test type: Superiority or Other; p = 0.321, Fisher Exact

ADVERSE EVENTS:
Arm/Group | AIC246 (60 mg) | AIC246 (120 mg) | AIC246 (240 mg) | Placebo
All-Cause Mortality (participants affected / at risk) | 2/33 | 1/31 | 1/34 | 1/33
Serious Adverse Events (participants affected / at risk) | 13/33 | 15/31 | 12/34 | 16/33
Other Adverse Events (participants affected / at risk) | 31/33 | 29/31 | 34/34 | 33/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AIC246 (60 mg) (N=33) | AIC246 (120 mg) (N=31) | AIC246 (240 mg) (N=34) | Placebo (N=33)
Pneumonia (Infections and infestations) | 2 (2) | 2 (2) | 2 (2) | 0 (0)
Epstein-Barr Virus Infestcion (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cytomegalovirus Infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 2 (2)
Alcaligenes Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Clostridial Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Enterococcal Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Human Herpesvirus 6 Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia Primary Atypical (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pneumonia Respiratory Syncytial Viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Septic Shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device Related Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Enterobacter Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes Virus Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia Bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute Myeloid Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Leukaemia Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Acute Lymphocytic Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diffuse Large B-Cell Lymphoma Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myelodysplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute Myeloid Leukaemia (in Remission) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-Hodgkin's Lymphoma Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute Graft Versus Host Disease in Intestine (Immune system disorders) | 4 (4) | 0 (0) | 2 (2) | 2 (2)
Acute Graft Versus Host Disease in Liver (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Graft Versus Host Disease (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute Graft Versus Host Disease in Skin (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoglykaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 0 (0) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Transplant Failure (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Anginga Pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomitting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
General Physical Health Deterioration (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Generalised Oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Hepatic Enzyme Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Liver Function Test (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Staphylococcus Test Positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Loss of Consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Venoocclusive Liver Disease (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal Failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AIC246 (60 mg) (N=33) | AIC246 (120 mg) (N=31) | AIC246 (240 mg) (N=34) | Placebo (N=33)
Diarrhoea (Gastrointestinal disorders) | 9 (11) | 9 (11) | 11 (14) | 10 (13)
Nausea (Gastrointestinal disorders) | 7 (8) | 8 (16) | 7 (7) | 11 (11)
Vomitting (Gastrointestinal disorders) | 4 (4) | 10 (11) | 8 (8) | 4 (7)
Constipation (Gastrointestinal disorders) | 4 (5) | 3 (3) | 3 (3) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 3 (3) | 3 (3) | 3 (3) | 5 (6)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 2 (3) | 4 (4) | 1 (1)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (1) | 2 (2) | 4 (4) | 2 (2)
Abdominal Distension (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (3) | 0 (0)
Abdominal Discomfort (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Dry Mouth (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 4 (4)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Anorectal Discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breath Odour (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colitis Ischaemic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Lip Dry (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Lip Swelling (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lip Ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral Discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Swollen Tongue (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gingivitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cytomegalovirus Infection (Infections and infestations) | 6 (6) | 6 (6) | 5 (5) | 11 (11)
Candidiasis (Infections and infestations) | 4 (4) | 1 (1) | 1 (1) | 3 (3)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 2 (2) | 2 (2) | 1 (1) | 2 (2)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 2 (2)
Eppstein-Barr Virus Infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Pseudomonas Infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 2 (2)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Oral Infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Respiratory Tract Infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Staphylococcal Infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Urinary Tract Infection Enterococcal (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Eppstein-Barr Viraemia (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Alcaligenes Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bacterial Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BK Virus Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Body Tinea (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clostridial Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cystitis Viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Enterococcal Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes Simplex (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Human Herpesvirus 6 Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Klebsiella Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Micrococcus Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oesphageal Candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral Candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral Herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Parainfluenzae Virus Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia Herpes Viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia Primary Atypical (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pneumonia Respiratory Syncytial Viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Septic Shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stenotrophomonas Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adenovirus Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cytomegalovirus Viraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Device Related Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Enterobacter Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fungal Skin Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes Virus Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Parotitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia Bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 4 (5) | 5 (7) | 4 (6) | 6 (7)
Puritus (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (4) | 5 (5) | 3 (4)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (5) | 4 (8) | 2 (2)
Dry Skin (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 1 (1) | 2 (2)
Rash Erythematous (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 1 (2) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Night Sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Rash Pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Actinic Keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute Febrile Neutrophilic Dermatosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermal Cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia Facial (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lichenfication (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nail Disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palmar Eythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Perivascular Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritis Generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rash Morbilliform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash Papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin Discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin Ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 3 (6) | 8 (9) | 4 (6) | 5 (5)
Oedema Peripheral (General disorders) | 4 (4) | 3 (3) | 8 (8) | 3 (3)
Pyrexia (General disorders) | 3 (3) | 4 (4) | 5 (5) | 6 (6)
Oedema (General disorders) | 1 (1) | 3 (3) | 2 (2) | 0 (0)
Chills (General disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Asthenia (General disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Catheter Site Erythema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Catheter Site Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Face Oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Local Swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Non-Cardiac Chest Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Application Site Hypersensitivity (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Axillary Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gait Distrubance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased Appetite (Metabolism and nutrition disorders) | 4 (4) | 2 (2) | 5 (5) | 3 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 4 (4) | 2 (2) | 2 (2) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 3 (3) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 2 (2) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Diabetes Mellitus (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Electrolyte Imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fluid Overload (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fluid Retention (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Food Intolerance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemosiderosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vitamin D Deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 8 (11) | 5 (5) | 1 (1)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 3 (3) | 1 (1) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 3 (3) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 3 (3) | 1 (1)
Lung Infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Postnasal Drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pulmonary Ebolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Bronchial Obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung Disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Painful Respiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngeal Erythema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory Disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Choking (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 4 (4) | 3 (3) | 8 (8) | 3 (3)
Neuropathy Peripheral (Nervous system disorders) | 3 (3) | 3 (3) | 1 (1) | 2 (2)
Tremor (Nervous system disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Polyneuropathy (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Burning Sensation (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypoaestesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Loss of Consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nystagmus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Restless Leg Syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ageusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Balance Disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VIIth Nerve Paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4) | 2 (3) | 1 (1)
Muscles Spasms (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (2) | 4 (6) | 0 (0)
Bone Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1) | 1 (1) | 2 (2)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 1 (1) | 1 (1)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Myopathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Arthrophathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Chest Wall Mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Exostosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle Atrophy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myosclerosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic Enzyme Increased (Investigations) | 2 (2) | 2 (2) | 1 (1) | 2 (2)
Blood Creatinine Increased (Investigations) | 1 (1) | 1 (3) | 1 (1) | 3 (3)
Alanine Aminotransferase Increased (Investigations) | 1 (1) | 0 (0) | 2 (3) | 1 (1)
Aspartate Aminotransferase Increased (Investigations) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Blood Alkaline Phosphatase Increased (Investigations) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Blood Folate Decreased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Blood Urea Increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Red Blood Cell Morphology Abnormal (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Transaminases Increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Weight Decreased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Blood Creatine Increased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Liver Function Test (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Antithrombin III Decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspergillus Test Positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood Amylase Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood Fibrinogen Decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood Potassium Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood Testosterone Decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
C-Reactive Protein Increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Computerised Tomogram Abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cytomegalovirus Test Positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Electrocardiogram QT Prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram ST Segment Elevation (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epstein-Barr Virus Test Positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gamma-Glutamyltransferase Increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lipase Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Polyomavirus Test Positive (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
White Blood Cell Count Decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Staphylococcus Test Positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute Graft Versus Host Disease (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Renal Failure (Renal and urinary disorders) | 5 (5) | 5 (5) | 3 (3) | 2 (2)
Nocturia (Renal and urinary disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Micturition Urgency (Renal and urinary disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Inconinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal Failure Acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Bladder Spasm (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry Eye (Eye disorders) | 1 (1) | 2 (2) | 5 (5) | 1 (1)
Conjunctivitis (Eye disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Vision Blurred (Eye disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (2)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Eye Irritation (Eye disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Lacrimation Increased (Eye disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Conjuctival Hyperaemia (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Eylid Oedema (Eye disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Eye Discharge (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye Pruritus (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Acute Graft Versus Host Disease in Skin (Immune system disorders) | 3 (4) | 5 (7) | 6 (7) | 2 (3)
Acute Graft Versus Host Disease in Intestine (Immune system disorders) | 3 (3) | 0 (0) | 5 (6) | 4 (5)
Graft Versus Host Disease (Immune system disorders) | 1 (1) | 2 (3) | 2 (2) | 0 (0)
Acute Graft Versus Host Disease in Liver (Immune system disorders) | 2 (2) | 0 (0) | 2 (2) | 3 (3)
Drug Hypersensitivity (Immune system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Chronic Graft Versus Host Disease (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seasonal Allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Ocular Discomfort (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sicca Syndrome (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Visual Impairment (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lagophthalmos (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 3 (5) | 2 (2) | 4 (4) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 2 (2) | 3 (3) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Splenomegaly (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Eosinophilia (Blood and lymphatic system disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Monocytosis (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymph Node Pain (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 5 (5) | 4 (4) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 3 (3) | 2 (2) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Psychotic Disorder (Psychiatric disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Decreased Activitiy (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mood Swings (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Panick Attack (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stress (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Adjustment Disorders (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fear (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Libido Decreased (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin Laceration (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Limb Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural Pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Scratch (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Suture Related Complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 2 (2) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 3 (3) | 2 (2)
Circulatory Collapse (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deep Vain Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hot Flush (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Orthostatic Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ischaemia (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Varicophlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute Myeloid Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Leukaemia Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Myelodysplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Acute Lymphocytic Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diffuse Large B-Cell Lymphoma Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Melanocytic Naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Multiple Myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute Myeloid Leukaemia (in Remission) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epstein-Barr Virus Associated Lymphoproliferative Disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Angina Pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pericardial Effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vulvovaginal Dryness (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Vulvovaginal Pruritus (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Atropic Vulvovaginitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspareunia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erectile Dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Genital Lesion (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Scrotal Erythema (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vaginal Discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast Pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast Swelling (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Venoocclusive Liver Disease (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cushingoid (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperparathyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Inappropriate Antidiuretic Hormone Secretion (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thyroid Disorder (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Auricular Swelling (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Middle Ear Effusion (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear Congestion (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear Pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Inner Ear Inflammation (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chimerism (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Every Publication, disclosure or other use of Information conveyed to the Institution and the Investigator in relation to the Trial and of data and results derived from the Performance of the Trial requires the express written consent of Sponsor.